# A double-blind, randomized, sham-controlled, exploratory trial of immunoadsorption in patients with chronic fatigue syndrome (CFS) including patients with Post-acute COVID-19 CFS (PACS-CFS)

# **Statistical Analysis Plan**

Version 2, of November 26, 2025

| Investigational medicinal pro | oduct: | Therapeutic | apheresis | with |
|-------------------------------|--------|-------------|-----------|------|
| immunoadsorption | | | | |

**Comparator**: sham Immunoadsorbtion (IA) (apheresis unit with a pre-saturated adsorber with immunoglobulins)

Indication: Post-COVID ME/CFS and ME/CFS

Sponsor: Charité Universitätsmedizin Berlin, Charitéplatz 1, 10117 Berlin

Financial support: Bfarm, Miltenyi

Alice Schneider, Deputy Statistician

Approved by

**Study registry identification**: ClinicalTrials.gov ID NCT05710770 **Development phase**: Post-Marketing (Exploratory), Phase IV

| Harald Prüß, Principal Investigator | |
|-------------------------------------|------------------------|
| | Place, Date, Signature |
| Friederike Ufer, Investigator | |
| | Place, Date, Signature |
| Ulrike Grittner, Statistician | |
| Chine Charlet, Stationelar | Place, Date, Signature |

Place, Date, Signature

# **Table of contents**

| 1 | Abbreviations | 3 |
|-------------|------------------------------------------|----|
| 2 | Background | 5 |
| 3 | Trial objective | 5 |
| 4 | Trial design | 5 |
| 4.1 | Inclusion and exclusion criteria | 11 |
| 4.2 | Power consideration | 13 |
| 5 | Analysis sets | 14 |
| 5.1 | Definitions | 14 |
| 5.2 | Application | 14 |
| 6 | Trial centres | 14 |
| 7 | Analysis variables | 14 |
| 7.1 | Demography and baseline characteristics | 15 |
| 7.2 | Primary variable | 16 |
| 7.3 | Secondary variables | 16 |
| 8 | Handling of missing values | 23 |
| 9 | Statistical analyses / methods | 23 |
| 9.1 | Demography and baseline characteristics | 23 |
| 9.2 | Primary analysis | 23 |
| 9.3 | Secondary analyses | 23 |
| 9.4 | Safety Analysis | 24 |
| 9.5 | Planned subgroup analyses | 24 |
| 10 | Interim analysis | 26 |
| 11 | Software | 26 |
| 12 | List of Changes in Version 2 of this SAP | 26 |
| 13 | References | 26 |
| 14 | Appendices | 29 |
| - ·<br>14.1 | • • | |
| 9.1 | | |
| 14.2 | | 31 |
| 14.3 | · | |
| 14.4 | e i | |

# 1 Abbreviations

| Abbreviation or special term | Explanation |
|---|---|
| ADA | anti-drug antibody |
| ADE | adverse device effect |
| AE | adverse event |
| ALT | alanine aminotransferase/transaminase |
| AST | aspartate aminotransferase/transaminase |
| BMI | Body Mass Index |
| BP | blood pressure |
| BVMT-R | Brief Visuospatial Memory Test - Revised |
| CCC 2003 | Canadian Consensus Criteria 2003 |
| CFS | chronic fatigue syndrome |
| CI | confidence interval |
| CRO | Contract Research Organisation |
| CRP | C-reactive protein |
| CSF | cerebrospinal fluid |
| DNA | deoxyribonucleic acid |
| EAS | effectiveness analysis set |
| ECG | electrocardiogram |
| EMG | electromyogram |
| EOS | end-of-study visit |
| EOT | end-of-treatment visit |
| eCRF | electronic Case Report Form |
| FAS | full analysis set |
| FAZ | Foveal Ávascular Zone |
| FDA | United States Food and Drug Administration |
| GCP | Good Clinical Practice |
| GCIPL | Ganglion Cell-Inner Plexiform Layer |
| IA | Immunoadsorption |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IP | Investigational Product |
| LPS 50+ | Leistungsprüfungssystem (performance testing system) for 50 to 90 years old |
| mITT | modified intention-to-treat set |
| MBL | mannose binding lectin |
| ME | myalgic encephalomyelitis |
| MoCA | Montreal Cognitive Assessment |
| NFL | neurofilament |
| OCB | oligoclonal IgG bands |
| OCT | Optical coherence tomography |
| PACS-CFS | Post-acute COVID-19 chronic fatigue syndrome |
| PBMC | peripheral blood mononuclear cells |
| PEM | post exertional malaise |
| PI | Principal Investigator |
| POTS | Postural Tachycardia Syndrome |
| PPS | per-protocol set |
| PR | pulse rate |
| PROMIS | patient-reported outcomes for health-related quality of life |

| pRNFL | peripapillary Retinal Nerve Fiber Layer |
|---|---|
| Qalb | CSF/serum quotient of total albumine |
| QoL | quality of life |
| RWT | Regensburger Wortflüssigkeits-Test (Regensburg Word Fluency Test) |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | Safety analysis set |
| SDMT | Symbol Digit Modalities Test |
| SoA | schedule of assessments |
| TAP | Test of attentional performance |
| Temp | body temperature (tympanic) |
| TMT-A / B | Trail Making Test A / B |
| TSH | thyroid-stimulating hormone |
| ULN | upper limit of normal |
| VLMT | verbal learning and memory test |
| WAIS-IV | Wechsler adult intelligence scale |
| WST | Wortschatz-Test (Vocabulary test) |

# 2 Background

There is an accumulation of evidence that a post-viral autoimmune reaction with the presence of autoantibodies targeting different neuronal tissues is involved in the pathogenesis of CFS/ME. Similarly, elevations of neurotransmitter receptor antibodies in patients with PACS- CFS have been observed. Furthermore, IA has shown clinical improvement in various types of autoimmune diseases associated with autoantibodies. Based on these findings, immunoadsorption may offer an effective treatment option for patients with CFS/ME, including patients with PACS-CFS. Results from first small studies indicate a beneficial therapeutic effect of IA in patients suffering from CFS/ME (Scheibenbogen et al., 2018; Tölle et al., 2020).

However, placebo-controlled trials investigating the effectiveness of IA in patients suffering from CFS/ME, including patients with PACS-CFS are lacking, although the procedure is generally well tolerated and safe. Having in mind the current number of confirmed COVID-19 cases, we might be facing a huge number of chronically ill severely disabled patients in the near future, underlining the ethical and economic urgency to develop effective therapeutic options for this devastating condition. Already before the association of the pandemic with a possible large outbreak of the disease became evident, an EU resolution from June 2020 indicated that more research is needed into this complex illness, supporting projects focusing on diagnostic tests and treatment in CFS/ME including PACS-CFS.

# 3 Trial objective

Due to the high number of patients suffering from CFS/ME, including PACS-CFS, the huge economic burden related to it, and the profound impairment of affected patients, there is an immense medical need to effectively treat patients with CFS/ME, including PACS-CFS. Therefore, in the present RCT, the effect of IA will be examined for the treatment of CFS/ME. Based on the assumed autoimmune pathogenesis underlying severe CFS/ME, it is tempting to hypothesize that this patient population will show clinical improvement (measured by the chalder fatigue score) after five treatments with immunoadsorption.

# 4 Trial design

This is a double-blinded, randomized, sham-controlled post-marketing (exploratory) trial to evaluate the therapeutic effect of five cycles of immunoadsorption every other day in 66 patients with CFS/ME, including patients with PACS-CFS. Two patient groups will be included (2:1), one receiving IA, one receiving a sham-apheresis.

A screening visit is planned up to max. 3 weeks (Day -42 to Day -21) before enrolment in the study to screen patients for eligibility (including blood and urine samples for safety parameters such as viral serology, pregnancy, drug and alcohol tests) and to assess demographics and medical history (table 1). In addition, cerebrospinal fluid and blood samples are taken to test for autoantibodies and markers of neurodegeneration or neuroinflammation. If a lumbar puncture was performed as part of the clinical routine within 6 months prior to the screening visit, it will not be repeated at screening. Patient reported outcome measurements such as Chalder Fatigue Scale, physical and autonomic function, quality of life and (in case of PACS-CFS) Post-COVID-19 Functional Status Scale questionnaires as well as Cognitive (MoCA and SDMT), physical (hand grip strength evaluation, 6MWT), and autonomic (Schellong-Test) assessments are performed at

screening or baseline visit. At baseline visit a detailed neuropsychological examination, and an assessment of physical function will be conducted.

Baseline assessments will be performed between Day -20 and -1 and in any case before the first IA cycle. These include a general and neurological physical examination assessing vital signs, ECG, body weight, repeating safety check for pregnancy. Blood samples for chemistry, hematology, coagulation and immunoglobulin titers are taken.

Patients are randomized either on Day -1 or Day 1 and a peripheral venous access (or Shaldon catheter) is implemented before the first IA cycle on Day 1 or Day 2 (Figure 1). Patients will be hospitalized at the clinical site from Day 1 to Day 9 or Day 10 and receive five IA treatments and medical visits including monitoring of coagulation every other day (i.e., on Days 1, 3, 5, 7, and 9 OR on Days 2, 4, 6, 8, and 10). If delays occur, the option to extend the in-hospital stay is available. Immunoadsorption can be postponed by one or more days.. Daily study nurse visits are scheduled including control of vital signs as well as questioning for AE(s).

After the last IA cycle, a blood sample for immunoglobulin titers is collected, the peripheral venous access (or Shaldon catheter) is removed and patients are discharged from the hospital if the investigator has no concerns. At EOT visit, patients will also complete the Chalder Fatigue Scale (Chalder et al., 1993), Fluge Score (Fluge et al., 2011; Fluge et al., 2015), and PEM questionnaires. In addition, patients will be instructed how to complete all of the requested questionnaires at home at follow up time points. If the IA treatments are performed according to the planned schedule, the end of treatment visit (EOT) will take place on Day 10. However, the EOT visit may vary between Day 9 and 12. If treatment needs to be terminated, the EOT can occur as early as day 2. In such cases, all examinations originally scheduled for day 10 will be conducted on the corresponding day. In addition, two of the four follow-up visits scheduled at month 2 (Day 60) and month 6 (Day 180; EOS, End of Study visit) will take place at the neurological wards and outpatient clinics respectively. Patients will be asked to bring all requested questionnaires (including Chalder Fatigue Scale), which they completed at home, to both follow-up visits, where further assessments and laboratory tests will be conducted. An optional second cerebrospinal fluid sample may also be taken on Day 60. The remaining two follow-up visits, scheduled at month 1 (Day 30) and month 4 (Day 120), will be conducted via telephone. During these visits, patients will be asked about any adverse events (AEs), concomitant medications, and questionnaires.

Immunoadsorption

Sham-apheresis

EOT

Follow-up

Sham-apheresis

Eos

Inpatient stay

Figure 1 Schematic illustration of the study design

Screening

BL

**Outpatient visits** 

Table 1: Schedule of Assessments

| Period/Visit name | SCR | BL <sup>6)</sup> | Treatment period (inpatient) | | | | | | | | | Follow-up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| renou/visit name | John | | | | | | | | | | EOT | US | | | | EOS |
| Study Days | -42 to -21 | -20 to -1 | 1 | 2 <sup>8)</sup> | 3 <sup>8)</sup> | 4 <sup>8)</sup> | 5 <sup>8)</sup> | 6 <sup>8)</sup> | <b>7</b> <sup>8)</sup> | 8 <sup>8)</sup> | 9-12 <sup>8)</sup> | | 30* <sup>6)</sup> | 60 <sup>6)</sup> | 120* <sup>6)</sup> | 180 <sup>6)</sup> |
| Time windows (days) | | | | | | | | | | | | | +/- 7 | +/- 7 | +/- 7 | +/- 7 |
| Status | | | | | | | | | | | | | | | | |
| Admission to hospital | | | Х | | | | | | | | | | | | | |
| Discharge from hospital | | | | | | | | | | | Х | | | | | |
| Discharge from study | | | | | | | | | | | | | | | | X |
| History | | | | | | | | | | | | | | | | |
| Informed consent | Х | | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | Χ | | | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | | | |
| Medical & Medication History | Х | | | | | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | | | | |
| Neurologic and general physical examination | Х | Х | | | | | | | | | Х | | | Х | | Х |
| Electrocardiogram (ECG) | Х | Х | | | | | | | | | Х | | | | | |
| Vital signs (BP, PR, and Temp) | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | | | | | Х |
| Body height | Х | | | | | | | | | | | | | | | |
| Body weight, BMI | Х | | | | | | | | | | Х | | | Х | | Х |
| Blood pregnancy | Х | Х | | | | | | | | | | | | | | |
| Urine test (dip sticks, drugs), alcohol test | Х | | | | | | | | | | | | | | | |
| Blood samples for chemistry, hematology | X <sup>(5)</sup> | Х | | | | | | | | | Х | | | Х | | Х |
| Thyroid hormone (TSH) | Х | | | | | | | | | | | | | | | |
| QuantiFERON ®-TB-Gold Plus-<br>Test <sup>5)</sup> and Viral Serologies <sup>5)</sup> | Х | | | | | | | | | | | | | | | |

\_\_\_\_\_

| Period/Visit name | SCR | BL <sup>6)</sup> | | Treatment period (inpatient) EOT US | | | | | | | | | | Follow-up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| T Grida, viole riamo | | | EOT | | | | | | | | | | | | | EOS |
| Study Days | -42 to -21 | -20 to -1 | 1 | 2 <sup>8)</sup> | 3 <sup>8)</sup> | 4 <sup>8)</sup> | 5 <sup>8)</sup> | 6 <sup>8)</sup> | 7 <sup>8)</sup> | 8 <sup>8)</sup> | 9-12 <sup>8)</sup> | | 30* <sup>6)</sup> | 60 <sup>6)</sup> | 120 <sup>*6)</sup> | 180 <sup>6)</sup> |
| Time windows (days) | | | | | | | | | | | | | +/- 7 | +/- 7 | +/- 7 | +/- 7 |
| Safety Assessments (cont.) | | | | | | | | | | | | | | | | |
| Blood samples for monitoring of coagulation | X <sup>(5)</sup> | х | | | | • | | | | | Х | | | Х | | |
| Monitoring of IA (IgG) | | | | | Before | e each a | nd after | last IA tr | eatment | | • | | | | | |
| Blood samples for immunoglobulin titers (IgA, IgG, IgM) | | Х | | | | | | | | | Х | | | Х | | Х |
| Adverse event questioning | | X | < | | | | | | | | | | | | | > |
| Concomitant Medications | | Х | < | | | | | | | | | | | | | > |
| Procedures | | | | | | | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | | | | | |
| PVA or Shaldon catheter implementation | | | 7 | X | | | | | | | | | | | | |
| Chest X-ray after Shaldon catheter implementation (if applicable) | | | 2 | X | | | | | | | | | | | | |
| Cranial MRI | | X <sup>9)</sup> | | | | | | | | | | | | Х | | |
| TheraSorb - Ig omni 5 adsorber cycles (IA active or IA sham) | | | | | 5 I | A treatm | nents eve | ery other | day | 1 | | | | | | |
| OCT | | Х | | | | | | | | | | | | Х | | |
| Removal of Shaldon catheter after last IA cycle | | | | | | | | | | | Х | | | | | |
| Lumbar puncture samples <sup>5)</sup> | Х | | | | | | | | | | | | | X <sup>3)</sup> | | |
| Blood samples for: - autoantibodies <sup>5</sup> - inflammatory markers (CRP, Ferritin, MBL, C3, C4), LDH, ACE - SARS-CoV-2 antibody-status | х | | | | | | | | | | | | | х | | х |
| SARS-CoV-2 PCR from nasopharyngeal swab | Х | Х | | | | | | | | | | | | | | |
| SARS-CoV-2 Antigen rapid test | | , | | | | | As requ | ired by o | current ho | ospital re | egulations | , | | | | |

| David dollait warea | SCR | BL <sup>6)</sup> | Treatment period (inpatient) | | | | | | | | | Follow-up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period/Visit name | JUN | DL. | EOT | | | | | | | EOT | T US | | | EOS | |
| Study Days | -42 to -21 | -20 to -1 | 1 | 2 <sup>8)</sup> | 3 <sup>8)</sup> | 4 <sup>8)</sup> | 5 <sup>8)</sup> | 6 <sup>8)</sup> | <b>7</b> <sup>8)</sup> | 8 <sup>8)</sup> | 9-12 <sup>8)</sup> | 30* <sup>6)</sup> | 60 <sup>6)</sup> | 120 <sup>*6)</sup> | 180 <sup>6)</sup> |
| Time windows (days) | | | | | | | | | | | | +/- 7 | +/- 7 | +/- 7 | +/- 7 |
| Questionnaires | | | | | | | | | | | | | | | |
| Chalder Fatigue Scale | X <sup>4)</sup> | | | | | | | | | | Х | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Fluge Score | | X <sup>4)</sup> | | | | | | | | | | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Assessment of post exertional malaise | | X <sup>4)</sup> | | | | | | | | | Х | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Bell Score | X <sup>4)</sup> | | | | | | | | | | Х | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Quality of life assessment (PROMIS) | | X <sup>4)</sup> | | | | | | | | | | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Physical function SF-36 | | X <sup>4)</sup> | | | | | | | | | Х | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Post-COVID-19 Functional Status<br>Scale (PACS- CFS patients only) | | X <sup>4)</sup> | | | | | | | | | | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| COMPASS-31 | | X <sup>4)</sup> | | | | | | | | | | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> | X <sup>4)</sup> |
| Physical assessment (-), hand grip strength) | Х | | | | | | | | | | Х | | Х | | X <sup>3)</sup> |
| 6 Minute Walking Test (6MWT) | | Х | | | | | | | | | | | Х | | |
| Schellong Test | | Х | | | | | | | | | Х | | Х | | X <sup>3</sup> |
| Detailed neuropsychiatric<br>examination (optional), VLMT,<br>BMVT-R, WAIS-IV, TAP, LPS 50+,<br>TMT-A / B, RWT, WST | | Х | | | | | | | | | | | х | | |
| Cognitive assessment (MoCA, PROMIS Cognitive Function Short Form 4a, SDMT) | | Х | | | | | | | | | | | Х | | |

Abbreviations: BMI = Body Mass Index [kg/m2]; BP = blood pressure; OCB = oligoclonal IgG bands; PR = pulse rate; CRP = C-reactive protein; MBL = Mannose binding lectin, Qalb = CSF/Serum quotient of total albumine; EOS = end-of-study visit; EOT = end-of-treatment visit; PBMC = Peripheral Blood Mononuclear Cells; PVA = Peripheral Venous Access; Temp. = body temperature (tympanic); TSH = Thyroid-stimulating hormone; US = unscheduled visit.

<sup>\*</sup>No on-site visit

<sup>&</sup>lt;sup>3)</sup>Only if requested by the investigator

<sup>&</sup>lt;sup>4)</sup> Completion by the patient at home

<sup>5)</sup> If not available in the 6 months prior to screening

\_\_\_\_\_

<sup>&</sup>lt;sup>6)</sup> Assessments can be done on several days; site personnel will schedule appointments with patients

<sup>7)</sup> In case of using results of lumbar puncture from clinical routine (up to 6 months prior to screening) these parameters cannot be collected at screening or baseline and therefore do not fall under a protocol deviation

<sup>8)</sup> If EOT occurs either before or after day 9-12, any examinations that were originally scheduled to take place on days 9-12, will be rescheduled to coincide with EOT that was determined at the time

<sup>&</sup>lt;sup>9)</sup> at day -60 to -1

# 4.1 Inclusion and exclusion criteria

Table 2: Inclusion Criteria

| Nr. | Inclusion Criterion | Variable | Values |
|---|---|---|---|
| 1 | Male and female subjects ≥18 years and < 65 years at time of informed consent | inex_0020 | yes/no |
| 2 | Body weight of ≥ 45 kilograms (kg) and ≤100 kg and must have a body mass index (BMI) within the range of 16-39.9 kg/m².at screening. BMI is calculated as Body weight (kg) / [Height (m)]² | inex_0030 | yes/no |
| 3 | Signed and dated informed consent prior to any study-mandated procedure | inex_0040 | yes/no |
| 4 | Chronic fatigue determined by the Chalder Fatigue Scale at screening | inex_0050 | yes/no |
| 5 | Diagnosis of chronic fatigue syndrome /myalgic encephalomyelitis (CFS/ME) under the 2003 Canadian Consensus Criteria (CCC) for ME/CFS syndrome and prolonged post-exertional malaise (PEM) including patients with CFS/ME due to Covid-19 (PACS-CFS) at screening. These criteria will be assessed by obtaining clinical histories and using appropriate symptom checklists. | inex_0060 | yes/no |
| 6 | Bell Score ≥ 20 and ≤ 50 | inex_0070 | yes/no |

Table 3: Exclusion Criteria

| Nr. | Exclusion Criterion | Variable | Values |
|---|---|---|---|
| 1 | Severe arterial hypotension (systolic BP < 100 mmHg, diastolic BP < 60 mmHg) at screening | inex_0080 | yes/no |
| 2 | Moderate to severe renal insufficiency (e.g., estimated glomerular filtration rate < 40 mL/min/1.73 m2, calculated by the Cockcroft-Gault formula or similar equation) | inex_0090 | yes/no |
| 3 | Cardiac insufficiency with an LVEF lower than 40% and/or uncontrolled cardiac arrhythmia | inex_0100 | yes/no |
| 4 | Coronary heart disease | inex_0110 | yes/no |
| 5 | Currently medication with ACE inhibitors and unable to switch to<br>another antihypertensive drug class within 2 weeks prior to baseline<br>visit (treatment with ACE inhibitors not allowed within 24 hours prior<br>to immune adsorption) | inex_0120 | yes/no |
| 6 | Malignant disease within the last 5 years | inex_0130 | yes/no |
| 7 | Clinically meaningful laboratory abnormalities at screening that would affect subject safety, as determined and documented by the investigator including but not limited to: Abnormal hematology: Hemoglobin < 8.0 g/dL, White Blood Cells count < 2.5/nL or >12/nL, Platelet count < 100/nL | inex_0140 | yes/no |
| | Abnormal liver function tests: ASAT/ALAT > 3 x higher than upper limit of reference (ULN), GGT, alkaline phosphatase > 3 x ULN, | | |

| | Total bilirubin > 2.0 mg/dL or PT-INR > 1.5 Note: Any parameter exceeding the above defined ULN should be re-checked once more as soon as possible, and in each case, prior to enrollment/randomization, to rule out lab error. | | |
|---|---|---|---|
| 8 | Any comorbidity bearing risk that patient might not tolerate treatment as judged by investigator | inex_0150 | yes/no |
| 9 | Medical, psychiatric or other conditions rendering patient incapable to understand the patient information and to give informed consent and maintain compliance during the trial | inex_0160 | yes/no |
| 10 | Fatigue duration for more than 5 years | inex_0170 | yes/no |
| 11 | Patients unwilling to have pseudonymized data recorded, analyzed and anonymously published | inex_0180 | yes/no |
| 12 | Participation in another clinical interventional trial within the last 6 months (or five half- lives, if longer than 6 months) previous to informed consent | inex_0190 | yes/no |
| 13 | Any surgical procedure requiring general anesthesia within 3 months prior to screening, or planned elective surgery during the study | inex_0200 | yes/no |
| 14<br>15 | Inmates of prisons or patients in psychiatric wards, or other state institutions Employee of the Sponsor, investigator or study site | inex_0210<br>inex_0220 | yes/no |
| 16 | Patient unable or unwilling to comply with study restrictions or procedures as described in Section 4. | inex_0230 | yes/no |
| 17 | Patient with known substance abuse or drug dependence currently or within one year prior to study participation, excluding nicotine and caffeine. This is determined through clinical history at screening. | inex_0240 | yes/no |
| 18 | Acute critical illness (intubation, ongoing Intensive Care Unit stay at the point of study involvement) | inex_0250 | yes/no |
| 19 | Acute or severe psychiatric disease (such as dementia, eating disorders, major unstable depression, bipolar affective disorder, schizophrenia, somatization disorders). Note: Follow-up by professionals will be offered when indicated. | inex_0260 | yes/no |
| 20 | Presence of other conditions or differential diagnosis better explaining the symptoms of the patient then the suspected ME/CFS, i.e., neuroendocrine diseases (such as thyroiditis or diabetes) | inex_0270 | yes/no |
| 21 | Ongoing immunomodulatory or immunosuppressive therapy or prior treatment with Rituximab (anti-CD20- antibody). | inex_0280 | yes/no |
| 22 | Clinical conditions that prohibit transitory volume changes or loss of plasma constituents other than Ig (e.g., serum albumin, electrolytes), equivalent to a plasma loss of about 10% per 1-fold processed plasma patient volume. | inex_0290 | yes/no |
| 23 | Indications that prohibit anticoagulation using Heparin and/or Anticoagulant Citrate Dextrose (ACD-A) solutions | inex_0300 | yes/no |
| 24 | Severe Hypercoagulability | inex_0310 | yes/no |

| 25 | Infection requiring hospitalization or intravenous administration of antibiotics/antimycotics or disease requiring administration of antivirus drugs (e.g., herpes zoster) within 4 weeks before starting the study treatment. | inex_0320 | yes/no |
|---|---|---|---|
| 26 | Acute infection with Cytomegalie Virus (CMV) or Eppstein-Barr Virus (EBV) | inex_0330 | yes/no |
| 27 | History of tuberculosis or evidence of active tuberculosis infection (positive QuantiFERON®-TB Gold Test). | inex_0340 | yes/no |
| 28 | Tested positive for any of the following in the Screening Phase: Human Immunodeficiency Virus (HIV), hepatitis B virus surface antigen (HBs antigen), hepatitis B virus core antibody (HBc antibody), and hepatitis C virus. Note: Patients positive for anti-HBs after Hep B vaccination but negative for hBsAg and anti-HBc are eligible (Hepatitis B serology: Appendix II). | inex_0350 | yes/no |
| 29 | Positive SARS-CoV-2 PCR test result at screening or baseline visit | inex_0360 | yes/no |
| 30 | Severe immune deficiencies (e.g., AIDS) | inex_0370 | yes/no |
| 31 | Suspected allergies against camelid antibodies or agarose | inex_0380 | yes/no |
| 32 | Pregnancy or breastfeeding at screening | inex_0390 | yes/no |
| 33 | Vaccination with live vaccines within 12 weeks prior to randomization and during study participation until 12 weeks after completion of immunoadsorption treatment | inex_0400 | yes/no |
| 34 | Non-live vaccination including vaccination against SARS-CoV-2 within 2 weeks prior to randomization and during the IA treatment period. Note: During the follow-up period, vaccination against SARS-CoV-2 will be allowed if in line with local regulations and if there are no concerns by the investigator. | inex_0410 | yes/no |
| 35 | Positive serum alcohol test | inex_0420 | yes/no |
| 36 | Positive test for drugs of abuse as per local standard at screening. | inex_0430 | yes/no |
| 37 | Donation of blood over 500 mL or 200 mL of plasma within 3 months prior to screening | inex_0440 | yes/no |
| 38 | Patient who has previously participated in this study and completed IA treatment | inex_0450 | yes/no |
| 39 | Any comorbidity bearing risk that patient might not tolerate treatment as judged by investigator | inex_0460 | yes/no |

## 4.2 Power consideration

In this study, a total of 66 patients (allocated in a 2:1 ratio: immunoadsorption (IA) group: 44 patients vs. sham group: 22 patients) will be included. Limited data from 2 small pilot studies, investigating IA in 10 patients with CFS/ME, is available to date. Consequently, data is lacking about precise effects, clinical outcomes, and effect sizes in this group of patients.

The justification of the sample size is based on the primary endpoint (change from baseline of the Chalder Fatigue Scale). The Chalder Fatigue Scale measures fatigue in patients using the overall score (range from 0 to 33) derived from a questionnaire with 11 questions (each scored from 0 to 3, see (Cella & Chalder, 2010; Chalder et al., 1993) for more details). Based on Cella & Chalder 2010, the mean score in a population of patients

suffering from CFS is 24.4 (with a standard deviation of 5.8) and for a healthy sample a mean value of 14.2 (with a standard deviation of 4.6) was observed. A difference of 10 points cannot be expected in this study since only patients suffering from CFS are included. In the systematic review of Nordin et al. 2016 a minimal important difference for the global change ranges between 2.3 and 3.3.

In an earlier study (Cleare et al. 1999) examining the efficacy of various treatments for CFS/ME, the difference in means of the Chalder Fatigue Scale was 4.5 points (Likert score) between the active and the control group. However, no sham-controlled study evaluating the effect of IA on CFS/ME has been conducted so far, but first pilot studies suggest a positive effect of IA in patients with CFS/ME.

To explore the expected precision obtained from the planned study, the distance from the mean group difference of the primary endpoint (change from baseline in Chalder Fatigue Scale) to the limits is calculated using its 95% confidence interval (CI) and a common standard deviation of 5.8 as provided for patient with CFS/ME in (Cella & Chalder, 2010). Using these assumptions and the given group sample sizes of 44 patients and 22 patients, the distance from mean to the limits of the 95%-CI is 3.03 points in the Chalder Fatigue Scale. Assuming an expected drop-out rate of 20% (resulting in expected group sample sizes of 35 and 18 patients, respectively) the distance from the mean to the limits of the 95%-CI increases to 3.37 points in the Chalder Fatigue Scale.

## 5 Analysis sets

#### 5.1 Definitions

The modified **full analysis set (FAS)** consists of a modified intention-to-treat (mITT) population and will include all patients that were randomized and underwent at least one IA cycle (active or sham IA intervention).

The **per-protocol set (PPS)** comprises all subjects who completed five cycles of their assigned intervention (IA or sham IA) as planned and who completed the study without critical protocol deviations.

The **safety analysis set (SAS)** will include all patients that underwent at least one IA cycle (active or sham IA intervention). Patients will be analyzed according to the intervention they received.

## 5.2 Application

The primary analysis is performed using the full analysis set (FAS), including the estimated values from multiple imputations for missing values. An analysis of the primary outcome using the PPS is used as a sensitivity analysis. All safety analyses will be done using the SAS (Safety analysis set).

#### 6 Trial centres

This is a single centre study with 66 patients.

## 7 Analysis variables

# 7.1 Demography and baseline characteristics

The following variables are assessed at baseline as additional patient characteristics:

Table 4: Demography and baseline characteristics

| Characteristic | Variable | Values |
|---|---|---|
| demographics | | |
| Age at inclusion (years) | dm_0010 | number |
| sex | dm_0020 | male, female, diverse |
| Body weight (kg) | dm_0031 | number |
| Body height (cm) | dm_0032 | number |
| BMI (kg/m²) | dm_0033 | number |
| Employment status | dm_0040 | employed, self-employed, currently unable to work, pension, student, unknown |
| Educational achievement | dm_0050 | No school-leaving certificate, lower secondary school leaving certificate (Hauptschule), higher secondary school leaving certificate (Realschule), grammar school (Gymnasium), completed vocational training, degree of a university of applied sciences, University, unknown |
| Self-reported predominant race | dm_0061 /<br>dm_0062<br>(other<br>specified) | Caucasian, African, Asian, Unknown, Other, please specify |
| Medical history | | |
| Pre-existing diseases | mh_0010 | yes, no |
| Pre-existing diseases: chapter | mh_0021 | e.g. diseases of the circulatory system |
| Pre-existing diseases: group | mh_0022 | e.g. Pulmonary heart disease and Diseases of the pulmonary circulation |
| Pre-existing diseases: subgroup | mh_0023 | e.g. Pulmonary embolism |
| Pre-existing diseases: ICD-Code | mh_0024 | e.g. I26 |
| Pre-existing diseases: ICD-Description | mh_0026 | e.g. Pulmonary embolism |
| Concomitant medications | cm_0021-<br>cm_0026 | Anatomical, therapeutically, chemical, ATC Code, active substance |
| Smoking | | |
| Smoking status | mh_0051 | Current smoker, former smoker, never smoker, unknown |
| Years of smoking | mh_0052,<br>mh_0054 | |

| Type of smoking | mh_0056 | e-cigarette, cigarette, other, unknown |
|---|---|---|
| Number of cigarettes per day | mh_0058 | |
| Known allergies | mh_0071 | yes, no |
| Type of allergy | mh_0072-<br>mh_0083 | Pollen allergy, House dust mite allergy,<br>Animal allergy, Hives, Sun allergy, Cross<br>allergies, Insect venom allergy, Drug<br>allergy |
| Anamnesis of infections | | |
| SARS-Cov-2 diagnosis in connection to fatigue | imh_0011 | yes, no |
| Other infection in connection to fatigue | imh_0021 | yes, no |
| Date of onset fatigue | imh_0031 | |

# 7.2 Primary variable

The primary outcome variable is the Chalder Fatigue Scale (Chalder et al., 1993) (range 0-33) at day 60.

## 7.3 Secondary variables

#### Safety related endpoints:

Occurrence of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and discontinuation due to TEAEs

Assessment of physical examinations, laboratory parameters, vital signs, and ECGs

#### Clinical effectiveness related endpoints

- Chalder Fatigue Scale (Chalder et al., 1993) at End of Treatment (EOT) visit and at month 1, 4, and 6 after the completion of IA
- Post-COVID-19 Functional Status (PCFS) scale (Klok et al., 2020) at month 1, 2, 4, and 6 after IA completion (only in patients with PACS-CFS)
- the SF-36 physical domain (Ware & Sherbourne, 1992) at EOT visit and at month 1, 2, 4, and 6 after IA completion
- Fluge questionnaire (Fluge et al., 2011; Fluge et al., 2015) at month 1, 2, 4, and 6 after IA completion
- PEM frequency, strength and severity by PEM questionnaire (Cotler et al., 2018) at EOT visit and at month 1, 2, 4, and 6 after IA completion
- the Bell disabling scale (Bell, 1995) at EOT visit and at month 1, 2, 4, and 6 after IA completion
- the Compass-31 questionnaire (Sletten et al., 2012) at month 1, 2, 4, and 6 after IA completion
- Schellong Test (Fanciulli et al., 2019) at EOT visit and at month 2 and optional month
   6 after IA completion
- hand grip strength test, at EOT and at month 2 and optional at month 6 after IA completion
- the 6 Minute Walking Test (6 MWT) ("ATS statement: guidelines for the six-minute walk test," 2002) at month 2 after IA completion
- optional neuropsychiatric assessment at month 2 after IA completion

- neurocognitive assessments (MoCA and SDMT) (Nasreddine et al., 2005) (Strober et al., 2020) at month 2 after IA completion
- quality of life (QoL) determined by the PROMIS questionnaire at month 1, 2, 4 and 6 after IA completion (Cella et al., 2019; Yang et al., 2019)
- PROMIS cognitive function short form 4a
- VLMT (verbal learning and memory test) (Helmstaedter et al., 2001)
- BVMT-R (brief visuospatial memory test revised) (Benedict, 1997)
- WAIS-IV (Wechsler adult intelligence scale) (Wechsler, 2008)
- TAP (Test of attentional performance) (Zimmermann & Fimm, 2004)
- LPS 50+ (Leistungsprüfungssystem (performance testing system) for 50 to 90 years old) (Sturm et al., 2015)
- TMT-A / B, Trail Making Test A / B (Reitan & Wolfson, 1993)
- RWT, Regensburger Wortflüssigkeits-Test (Regensburg Word Fluency Test) (Aschenbrenner et al., 2000)
- WST, Wortschatz-Test (Vocabulary test) (Schmidt & Metzler, 1992)

## Biomarker related endpoints:

- biomarkers of autoimmune activity (autoantibody titers against neurotransmitter receptors; among others ß2-adeno-receptor- and muscarine- receptor-antibodies) in blood at month 2 and 6 and optional in cerebrospinal fluid at month 2 after IA completion
- immunostatus (differential blood, IgG, IgM, IgA fractions) in blood at EOT, at month 2 and 6 after IA completion
- immunoglobulin levels (including SARS-CoV-2 antibody titers and PCR, if applicable) at month 2 and 6 in blood and optional in cerebrospinal fluid at month 2 after IA completion
- inflammatory biomarkers in blood (CRP, ferritin, MBL, white blood cell count, complement factors, immunoglobulin level and subtype) at month 2 and 6 after IA completion
- autoantibodies against known or unknown neuronal epitopes (Stöcker- autoimmuneencephalitis panel and screening via immunofluorescent staining on mouse brain sections – in cooperation with separate project EA1/258/18) in blood and optional in cerebrospinal fluid after IA completion.
- neurofilament (NFL) in cerebrospinal fluid at month 2 after IA completion
- auto-antibody and vaccine titers in serum and cerebrospinal fluid as well as intrathecal synthesis (CFS) at month 2 after IA completion
- inflammatory biomarkers in cerebrospinal fluid (white cell count, total protein, CSF/serum quotients of albumin (Qalb), lactate, oligoclonal IgG bands (OCB), cytokines)) at month 2 after IA completion
- MRI parameter: grey matter volume, white matter volume, thalamus volume left and right, thalamic functional connectivity to sensomotoric cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, EndoPAT Reactive Hyperemia Index (RHI). Volumetry is based on a high-resolution T1-weighted MPRAGE sequence (voxel size 1 mm isotropic, FOV 256 mm, TR = 2500 ms, TE = 2.64 ms). The functional connectivity measures are derived from a BOLD-sensitive resting-state EPI sequence (720 volumes, voxel size 2 mm isotropic, TR = 800 ms, TE = 37 ms, FOV 208 mm).
- OCT parameter: ganglion cell-inner plexiform layer (GCIPL), peripapillary retinal nerve fiber layer (pRNFL), foveal avascular zone (FAZ), vessel density
- CD11c-Expression: Mean fluorescence intensity (MFI) on total CD19<sup>+</sup> B cells, Percentage of CD11c<sup>-</sup> cells within the CD19<sup>+</sup> gate, CD11c MFI and %CD11c<sup>-</sup> specifically on IgD<sup>-</sup>CD27<sup>+</sup> memory B cells (CD19<sup>+</sup>IgD<sup>-</sup>CD27<sup>+</sup> gate)
- IgM Expression: Mean fluorescence intensity (MFI) on total CD19<sup>+</sup> B cells, Percentage of IgM<sup>-</sup> cells within the CD19<sup>+</sup> gate, IgM MFI and %IgM<sup>-</sup> specifically on

IgD<sup>-</sup>CD27<sup>+</sup> memory B cells (CD19<sup>+</sup>IgD<sup>-</sup>CD27<sup>+</sup> gate), Activated Canonical Class-Switched Memory B Cells (aCSM), CD19<sup>+</sup>IgD<sup>-</sup>IgM<sup>-</sup>CD27<sup>+</sup>CD11c<sup>-</sup>, Frequency quantification within total B cells or parent gates, Activated canonical class-switched memory B cells

Table 5: primary and secondary outcome variables

| Characteristic | Variable | Values |
|---|---|---|
| Primary outcome variable | | |
| Chalder Fatigue Scale at 2 months | cfs_0001-cfs_0011 | 11 items with levels 0-3 each, sum score has to be calculated |
| Secondary outcome variables | | |
| Efficacy related outcomes | | |
| Chalder Fatigue Scale at<br>End of Treatment (EOT)<br>visit and at month 1, 2, 4,<br>and 6 after the completion<br>of IA | cfs_0001-cfs_0011 | 11 items with levels 0-3 each, sum score has to be calculated |
| Post-COVID-19<br>Functional Status (PCFS)<br>scale | pcfs_0020-pcfs_0050 | Ordinal scale, range 0 to 4 (0: no limitations, 4: severe limitations), |
| SF-36 physical domain Fluge questionnaire | sf_0041-sf_0050 ccc_0011-ccc_0131 | 10 items, each scored with: no limitations (0 points), some limitations (5 points), severe limitations (10points), the sum will be calculated 5 domains with different number of items, domains: fatigue, pain, cognition, circulation, each item is scored from 0 to 10 according to the severity (10: highest severity), domains will be analyzed separately |
| Post-Exertional Malaise (PEM) | pem_0021-pem_0110 | 11 items, 5 items<br>scored 0 to 4 for<br>frequency, 5 items<br>scored 0 to 4 for<br>severity, 1 item scored<br>0 to 6 for duration, sum<br>score from 0 to 46 |
| Bell Score | bell_0020 | 1 item with 11 statements, 0-100 |

| Compass-31 | com_0001-com_0031 | points (100: no symptoms, 0: severe symptoms) 31 items in 6 domains, score by domain are |
|---|---|---|
| | | score by domain are rescaled ranging from 0 to 100 |
| Schellong Test /POTS | pst_0021-pst_0080 | Using items to evaluate if POTS is present (Increase in heart rate within 10 minutes of standing by at least 30 beats/minute above the level when lying down or, to at least 120 beats/minute absolutely, no pathological drop in blood pressure (i.e., systolic drop not more than 20 mm Hg and diastolic drop not more than 10 mm Hg), increasing symptoms of orthostatic intolerance) |
| 6 Minute Walking Test (6 MWT) | | |
| MoCA | moca_0011-moca_0110 | Score items, sum of maximum 30 or 31 points dependent on educational level |
| Symbol Digit Modalities<br>Test, SDMT | sdmt_0020 | Item on number of correct remembered words after 90 seconds |
| PROMIS-29, physical function, anxiety, depression, pain interference, pain severity, fatigue, sleep disturbance, ability to participate in social roles and activities | pfa11-pfa53, edanx01-edanx53, eddep04-eddep41, hi7, an3, fatexp41, fatexp40, sleep109, sleep116, sleep20, sleep44, srpper11_caps-srpper46_caps, pain9-pain34, global07 | each of the 7 domains<br>will be scored<br>separately,<br>transformation in<br>standardized t-values |
| PROMIS cognitive function short form 4a | pc2r-pc42r | Sum score converted to t score |
| Additional secondary outcome variables | | |
| VLMT (verbal learning and memory test) | vlmt_0011 - vlmt_0220 | total score: addition of the learning achievements of the 5 |

| | | rounds; delayed recall: number of words correctly recalled from the word list after a time delay; loss after delay: subtraction of the number of correctly recalled words in learning session 7 from the number of correctly recalled words in learning session 5; correct recognition: subtraction of the number of false positives and interference items from the number of correctly recognised words in the first list (i.e.: 18. recognition performance (W) - (19. interference + 20. false positives)). |
|---|---|---|
| BVMT-R (brief visuospatial memory test revised) | bmvt_0011 — bmvt_0150 | total score: addition of the points from all three trials; delayed recall: number of correctly remembered figures. (correct figure and correct place); percent retained: [delayed recall / (higher of trial 2 and trial 3)] x 100; recognition discrimination index: (recognition hits) - (recognition false alarms) |
| WAIS-IV (Wechsler adult intelligence scale) | wais_0011 - wais_0070 | forward: number of correctly repeated number sequences; backwards: number of number sequences correctly recited backwards; sequential: number of correctly sequenced number sequences. |
| TAP (Test of attentional performance) | tap_0011 - tap_0100 | median of the reaction<br>time. (runs without<br>warning tone); standard<br>deviation of the reaction |

time. (runs without warning tone); number of omissions in the sustained attention task; number of omissions of auditory stimuli; number of omissions of visual stimuli. LPS 50+ number of correctly lps\_0010 - lps\_0040 (Leistungsprüfungssystem solved lines. (performance testing system) for 50 to 90 years old) TMT-A / B, Trail Making tmt\_0011 - tmt\_0060 number of seconds to Test A / B complete the task A; number of seconds to complete the task B; TMT B/A ratio = time TMT-A / time TMT-B number of animals or RWT, Regensburger rwt\_0011 - rwt\_0080 Wortflüssigkeits-Test first names mentioned within 60 seconds; (Regensburg Word Fluency Test) number of S-words or M-words mentioned within 60 seconds. WST, Wortschatz-Test wst 0010-wst 0050 raw score (sum of (Vocabulary test) correct values) Biomarker related endpoints biomarkers of stoe 0023-stoe 0025, ak 0011-ak 0063 autoimmune activity (autoantibody titers against neurotransmitter receptors; among others ß2-adeno-receptor- and muscarine- receptorantibodies), autoantibodies against known or unknown neuronal epitopes immunostatus (differential ig 0011-ig 0063 blood, IgG, IgM, IgA fractions) immunoglobulin levels inf 0121-inf 0140, imh 0011, imh 0012, ig 0011-(including SARS-CoV-2 ig 0023 antibody titers and PCR, if applicable)

| inflammatory biomarkers in blood (CPR) ferritin, MBL, white blood cell count, complement factors, immunoglobulin level and subtype) neurofilament (NFL) auto-antibody and vaccine titers in serum and cerebrospinal fluid as well as intrathecal synthesis (CFS) inflammatory biomarkers in serum and cerebrospinal fluid (white cell count, total protein, CSF/serum quotients of albumin (Calb), lactate, oligoclonal IgG bands (OCB), cytokines)) MRI measures: grey matter volume, white matter volume, thalamus volume left and right, thalamic functional connectivity to sensomotor cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional connectivity to visuo-occipital visus left and right, EndoPAT Reactive Hyperemia Index (RHII) OCT: ganglion cell-inner plexiform layer (GCIPL), peripapillary retinal nerve fiber layer (GRNFL), foveal avascular zone (FAZ), vessel density CD11c Expressions (CD19+ B cells, IgM Expressions, Activated canonical class-switched memory B cells witched memory B cells witched memory B cells switched memory B cells perc_cd11cp_l_dprincd27pl_cd19pl, perc_d11pl, perc_assm_lgdmin_cd27pl_cd11pl, perc_assm_lgdmin_cd27pl_cd11pl, perc_assm_lgdmin_cd27pl_cd11pl, perc_assm_lgdmin_cd27pl_cd19pl | | |
|---|---|---|
| auto-antibody and vaccine titers in serum and cerebrospinal fluid as well as intrathecal synthesis (CFS) inflammatory biomarkers in serum and cerebrospinal fluid (white cell count, total protein, CSF/serum quotients of albumin (Qalb), lactate, oligoclonal IgG bands (OCB), cytokines)) MRI measures: grey matter volume, white matter volume, thalamus volume left and right, thalamic functional connectivity to sensomotoric cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional replexiform layer (GCIPL), peripapillary retinal nerve fiber layer (pRNFL), foveal avascular zone (FAZ), vessel density CD11c Expressions (CD19+ B cells, IgD**CD27** memory B cells), IgM Expressions, Activated canonical class-switched memory B cells switched memory B cells switched memory B cells ak _0011-ak_0063 ak _0011-ak_0011 abem_0273, chem_0011- chem_0273, chem_0011- chem_0273, chem_0011- chem_0011- chem_00271, chem_0011- chem_00271, chem_0011- chem_00273, chem_0011- chem_00271, chem_0011- chem_00 | in blood (CRP, ferritin, MBL, white blood cell count, complement factors, immunoglobulin | inf_0161-inf_0173 |
| vaccine titers in serum and cerebrospinal fluid as well as intrathecal synthesis (CFS) inflammatory biomarkers in serum and cerebrospinal fluid (white cell count, total protein, CSF/serum quotients of albumin (Qalb), lactate, oligoclonal IgG bands (OCB), cytokines)) MRI measures: grey matter volume, thalamus volume left and right, thalamic functional connectivity to sensomotoric cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, thalamic functional connectivity to peripapillary retinal nere plexiform layer (GCIPL), peripapillary retinal nere plexiform layer (GCIPL), foveal avascular zone (FAZ), vessel density CD11c Expressions (CD19+ B cells, IgD*CD27* memory B cells), IgM Expressions, Activated canonical class-switched memory B cells switched memory B cells switched memory B cells switched memory B cells switched memory B cells perc_acsm_igdmin_cd27pl_cd19pl, perc_igmpl_cd11pl, perc_acsm_igdmin_cd27pl_cd11pl, perc_igmpl_cd11pl, perc_acsm_igdmin_cd27pl_cd11pl, perc_acsm_igdmin_cd27p | neurofilament (NFL) | liq_0161-liq_0163, liq_0171-liq_0173 |
| in serum and cerebrospinal fluid (white cell count, total protein, CSF/serum quotients of albumin (Qalb), lactate, oligoclonal IgG bands (OCB), cytokines)) MRI measures: grey matter volume, thalamus volume telf and right, thalamic functional connectivity to sensomotoric cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, EndoPAT Reactive Hyperemia Index (RHI) OCT: ganglion cell-inner plexiform layer (GCIPL), peripapillary retinal nerve fiber layer (pRNFL), foveal avascular zone (FAZ), vessel density CD11c Expressions (CD19+ B cells, IgM Expressions, Activated canonical class-switched memory B cells switched memory B cells switched memory B cells and replaced an | vaccine titers in serum<br>and cerebrospinal fluid as<br>well as intrathecal | ak_0011-ak_0063 |
| matter volume, white matter volume, thalamus volume left and right, thalamic functional connectivity to sensomotoric cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, EndoPAT Reactive Hyperemia Index (RHI) OCT: ganglion cell-inner plexiform layer (GCIPL), peripapillary retinal nerve fiber layer (pRNFL), foveal avascular zone (FAZ), vessel density CD11c Expressions (CD19+ B cells, IgD CD27+ memory B cells), IgM Expressions, Activated canonical class-switched memory B cells withalamus_r_volume, thalamic_motor_I_fc, thalamic_occipital_fc, th | in serum and cerebrospinal fluid (white cell count, total protein, CSF/serum quotients of albumin (Qalb), lactate, oligoclonal IgG bands | |
| plexiform layer (GCIPL), peripapillary retinal nerve fiber layer (pRNFL), foveal avascular zone (FAZ), vessel density CD11c Expressions (CD19+ B cells, IgD^CD27+ memory B cells), IgM Expressions, Activated canonical class- switched memory B cells Switched memory B cells plexiform layer (GCIPL), peripapillary retinal nerve fiber layer (pRNFL), foveal avascular zone (FAZ), vessel density z_cd11c_exp_cd19pl, perc_cd11cpl_cd27plus_cd19pl, perc_cd11cpl_igdmin_cd27pl_cd19pl, perc_igmpl_igdmin_cd27pl_cd19pl, perc_igmpl_igdmin_cd27pl_cd11cmin_cd 19pl, perc_cl_acsm_igdmin_cd27pl_cd19pl | matter volume, white matter volume, thalamus volume left and right, thalamic functional connectivity to sensomotoric cluster left and right, thalamic functional connectivity to visuo-occipital cluster left and right, EndoPAT Reactive Hyperemia | thalamus_r_ volume, thalamic_motor_lfc, thalamic_motor_rfc, thalamic_occiptial_lfc, |
| (CD19+ B cells, IgD-CD27+ memory B cells), IgM Expressions, Activated canonical class-switched memory B cells Switched memory B cells Z_cd11c_exp_igdmin_cd27plus_cd19pl, perc_cd11cpl_igdmin_cd27pl_cd19pl, z_igm_exp_cd19pl, perc_igmpl_igdmin_cd27pl_cd19pl, perc_igmpl_igdmin_cd27pl_cd11cmin_cd 19pl, perc_cl_acsm_igdmin_cd27pl_cd19pl | plexiform layer (GCIPL),<br>peripapillary retinal nerve<br>fiber layer (pRNFL),<br>foveal avascular zone | gcipl, prnfl, faz, vessel_density_full |
| Safety related endpoints | (CD19+ B cells,<br>IgD-CD27+ memory B<br>cells), IgM Expressions,<br>Activated canonical class- | z_cd11c_exp_igdmin_cd27plus_cd19pl, perc_cd11cpl_cd19pl, perc_cd11cpl_igdmin_cd27pl_cd19pl, z_igm_exp_cd19pl, z_igm_exp_igdmin_cd27pl_cd19pl, perc_igmpl_cd19pl, perc_igmpl_igdmin_cd27pl_cd19pl, perc_acsm_igdmin_igmmin_cd27pl_cd11cmin_cd |
| | Safety related endpoints | |

| Adverse events and | ae_0053, sae_0123 |
|-----------------------|-------------------|
| severe adverse events | |

## 8 Handling of missing values

Missing data will be categorized according to Rubin as "missing completely at random", "missing at random" and "missing not at random" (MCAR, MAR and MNAR) (RUBIN, 1976). For missing data in outcome variables, data will be imputed using multiple imputation by chained equations (mice) (Van Buuren & Van Buuren, 2012) with the R package MICE (van Buuren & Groothuis-Oudshoorn, 2011) with 30 imputed data sets, where appropriate is the assumption of MAR or MCAR is reasonable. It is planned to perform sensitivity analyses, in which the robustness of the inference will be investigated. Sensitivity analyses will be done using complete data without any imputation. The following variables will be used for the imputation process: all outcome variables, demographic variables age, sex, and BMI.

# 9 Statistical analyses / methods

## 9.1 Demography and baseline characteristics

Demography and baseline characteristics will be reported for the total population and by treatment arm using descriptive statistical summary measures. No statistical test will be performed to compare baseline characteristics between randomized treatment groups. For continuous variables, mean with standard deviation (SD), median, interquartile range (IQR), minimum, maximum will be given depending on the distribution of the respective characteristic. For categorical data absolute and relative frequencies are given for each category.

## 9.2 Primary analysis

For the primary outcome, the Chalder Fatigue Scale at 2 months, descriptive statistics will be presented for both treatment arms. This will include the number of participants (n), mean, standard deviation (SD), median, interquartile range (IQR), minimum, and maximum for the continuous total score. Additionally, for the categorical responses (e.g., presence/absence of fatigue), frequencies and percentages will be reported.

Confirmatory analysis of the primary outcome will be conducted based on the full analysis set. An analysis of covariance (ANCOVA) will be conducted. The dependent variable is the Chalder Fatigue Score at day 60, independent variables include baseline Chalder Fatigue Score, treatment group (intervention / control), and age at baseline. The effect estimate for the treatment variable and the corresponding 95%Cl will be reported. Sensitivity analysis will be done using the PPS without imputation of missing values.

#### 9.3 Secondary analyses

For all secondary endpoints, descriptive statistics will be calculated and presented at each time point of measurement for both treatment groups. For continuous secondary outcomes, this will include the mean, standard deviation, median, interquartile range, minimum, and maximum. For categorical or ordinal secondary outcomes, frequencies and percentages will be reported. These descriptive summaries will be presented in tabular format, and appropriate graphical representations, such as line plots for longitudinal data, bar charts, or box plots, will be utilized to visually depict trends, distributions, and differences between treatment arms across all assessment time points. For all secondary endpoints, analysis of

covariance (ANCOVA) models will be employed, analogous to the approach for the primary outcome. The choice of link function will be tailored to the specific nature of each outcome variable (e.g., linear for continuous outcomes, binary logistic for dichotomous outcomes, or ordinal for ordered categorical outcomes). In instances of repeated measures, mixed-effects regression models will be utilized, incorporating random intercepts for individual participants to account for within-subject correlation. Each model will include the respective baseline value of the endpoint, age at baseline, and treatment group as fixed effects. Effect estimates for the treatment variable, along with their 95% confidence intervals (CI), will be reported. All analyses will be conducted using the Full Analysis Set (FAS). Sensitivity analyses will be performed using the Per-Protocol Set (PPS), without imputation of missing values, to assess the robustness of the findings.

Responder analysis: Explorative analyses comparing responders and non-responders in both groups regarding PCS-associated signature at baseline: CD11c and IgM expression and an aCSM frequency. For this analysis a binary logistic regression model will be implemented with the responder (yes/no) variable as the dependent variable, the PCS-associated signature at baseline, the group and the interaction term between PCS-signature at baseline and group as independent variables.

# 9.4 Safety Analysis

Descriptive methods will be used for analysis of safety parameters, adverse events and their intensity in total and reported separately for the intervention groups. Incidence rates and 95% confidence intervals (CI) will be calculated using Poisson regression models that consider the different observation periods for each participant. Group comparisons will be made using incidence rate ratios and their 95% Cls. The safety analysis results will be carefully interpreted and discussed, even for minor group differences, as statistical significance is not the main focus in this context. A comprehensive listing of all individual patient adverse events (AEs) and severe adverse events (SAEs) will be presented. This will include, for each event, the patient identifier, treatment arm, AE/SAE term (coded using Medical Dictionary for Regulatory Activities [MedDRA]), verbatim term, onset date, resolution date, severity (e.g., mild, moderate, severe), seriousness criteria (if applicable), causality assessment (e.g., related, not related to study drug), action taken with study drug, and outcome. Separate listings will be generated for AEs and SAEs. Furthermore, any AEs leading to study drug discontinuation or study withdrawal will be specifically highlighted. These listings will serve as a detailed and transparent record for safety monitoring and will facilitate thorough review by medical monitors and regulatory authorities.

## 9.5 Planned subgroup analyses

For the statistical analyses of the subgroups, the models defined in the sections above will be used for the respective outcome, additionally with an interaction term of the treatment group variable with the subgroup, in order to obtain indications of differential treatment effects in the subgroups. We will report effect estimates of interaction effects with corresponding 95%CI. In addition, marginal effect estimates for each subgroup and 95% confidence intervals will be provided.

| Sub-group (levels) | Outcomes |
|---|---|
| Sex (male, female, diverse) | Primary endpoint and efficacy related secondary endpoints |
| <b>Age</b> (< 40 years, ≥ 40 years) | Primary endpoint and efficacy related secondary endpoints |

\_\_\_\_\_

| Sub-group (levels) | Outcomes |
|---|---|
| <b>Education</b> (higher education meaning A-levels or higher, medium or lower educational achievement) | Primary endpoint and efficacy related secondary endpoints |
| Employment status<br>(retired/ currently unable to<br>work, employed/ self-employed<br>/ student) | Primary endpoint and efficacy related secondary endpoints |
| <b>Body-mass index (BMI)</b> $(< 30 \text{ kg}^*\text{m}^{-2}, \ge 30 \text{ kg}^*\text{m}^{-2})$ | Primary endpoint and efficacy related secondary endpoints |
| ME/CFS vs. Post-COVID-<br>ME/CFS | Primary endpoint and efficacy related secondary endpoints, OCT outcome: Retinal vascular and perfusion density in the superficial vascular plexus (SVP) |
| Disease duration<br>(≤2.5 years, >2.5 years) | Primary endpoint and efficacy related secondary endpoints |
| Bell Score at baseline (≤30, >30) | Primary endpoint and efficacy related secondary endpoints |
| Chalder Fatigue Scale at baseline (≤20, >20) | Primary endpoint and efficacy related secondary endpoints |
| Focal neurological deficit at baseline (yes, no) | Primary endpoint and efficacy related secondary endpoints |
| Antineuronal autoantibodies (yes, no) | Primary endpoint and efficacy related secondary endpoints |
| Subgroups by 7 PROMIS 29 sub domains (T-score cut offs of 30-40) | Primary endpoint and efficacy related secondary endpoints |
| Baseline detection of<br>GPCR-Autoantibodies (pos.<br>result from Labor Celltrend;<br>yes, no) | Primary endpoint and efficacy related secondary endpoints |
| Subgroups by the presence of specific B-cell subpopulations at baseline (incl. activated plasma blasts, memory like and activated naïve like cells identified in CyTOF analysis) | Primary endpoint and efficacy related secondary endpoints |
| Subgroups by baseline retinal nerve fibre layer (pRNFL) thickness (median split) | Primary endpoint and efficacy related secondary endpoints |

| Sub-group (levels) | Outcomes |
|---|---|
| Subgroups by baseline retinal ganglion cell layer (GCIPL) thickness (median split) | Primary endpoint and efficacy related secondary endpoints |

# 10 Interim analysis

An interim analysis is not planned.

#### 11 Software

R (version 4.4.2 or later) will be used. For multiple imputation of missing values, the package mice will be used (van Buuren and Groothuis-Oudshoorn (2011)). For mixed models, the R package Ime4 will be used (Bates et al. (2015)). For marginal mean estimates, the R package emmeans will be used (Lenth (2024)).

# 12 List of Changes in Version 2 of this SAP

- MRI and OCT added in tables for scheduled measures
- MRI and OCT variables added in outcome and variable tables and listings,
- Additional immunological biomarkers: CD11c-Expression, IgM-Expression, Activated canonical class-switched memory B cells
- Additional subgroup analysis by OCT parameters (Subgroups by reduced peripapillary retinal nerve fibre layer, pRNFL/ganglion cells or inner plexiform layer; GCIPL at baseline)
- Additional OCT Outcome for subgroup analysis on subgroup defined by ME/CFS vs. Post-COVID-ME/CFS.
- Responder analysis in section 9.3: Explorative analyses comparing responders and non-responders in the intervention group regarding PCS-associated signature at baseline: CD11c and IgM expression and an aCSM frequency.

#### 13 References

- Aschenbrenner, S., Tucha, O., & Lange, K. W. (2000). *Regensburger wortflüssigkeits-test: RWT*. Hogrefe, Verlag für Psychologie.
- ATS statement: guidelines for the six-minute walk test. (2002). *Am J Respir Crit Care Med*, 166(1), 111–117. <a href="https://doi.org/10.1164/ajrccm.166.1.at1102">https://doi.org/10.1164/ajrccm.166.1.at1102</a>
- Bates, D., Mächler, M., Bolker, B., & Walker, S. (2015). Fitting Linear Mixed-Effects Models Using Ime4. *Journal of Statistical Software*, 67(1), 1 48. https://doi.org/10.18637/jss.v067.i01
- Bell, D. S. (1995). The doctor's guide to chronic fatigue syndrome: understanding, treating, and living with CFIDS. Addison-Wesley Pub. Co.
- Benedict, R. H. (1997). Brief visuospatial memory test--revised. PAR.
- Cella, D., Choi, S. W., Condon, D. M., Schalet, B., Hays, R. D., Rothrock, N. E., Yount, S., Cook, K. F., Gershon, R. C., Amtmann, D., DeWalt, D. A., Pilkonis, P. A., Stone, A. A., Weinfurt, K., & Reeve, B. B. (2019). PROMIS((R)) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. *Value Health*, 22(5), 537–544. https://doi.org/10.1016/j.jval.2019.02.004
- Cella, M., & Chalder, T. (2010). Measuring fatigue in clinical and community settings. *J Psychosom Res*, *69*(1), 17–22. <a href="https://doi.org/10.1016/j.jpsychores.2009.10.007">https://doi.org/10.1016/j.jpsychores.2009.10.007</a>

- Chalder, T., Berelowitz, G., Pawlikowska, T., Watts, L., Wessely, S., Wright, D., & Wallace, E. P. (1993). Development of a fatigue scale. *J Psychosom Res*, 37(2), 147–153. https://doi.org/10.1016/0022-3999(93)90081-p
- Cotler, J., Holtzman, C., Dudun, C., & Jason, L. A. (2018). A Brief Questionnaire to Assess Post-Exertional Malaise. *Diagnostics (Basel)*, 8(3). https://doi.org/10.3390/diagnostics8030066
- Fanciulli, A., Campese, N., & Wenning, G. K. (2019). The Schellong test: detecting orthostatic blood pressure and heart rate changes in German-speaking countries. *Clin Auton Res*, 29(4), 363–366. <a href="https://doi.org/10.1007/s10286-019-00619-7">https://doi.org/10.1007/s10286-019-00619-7</a>
- Fluge, O., Bruland, O., Risa, K., Storstein, A., Kristoffersen, E. K., Sapkota, D., Naess, H., Dahl, O., Nyland, H., & Mella, O. (2011). Benefit from B-lymphocyte depletion using the anti-CD20 antibody rituximab in chronic fatigue syndrome. A double-blind and placebo-controlled study. *PLoS One*, *6*(10), e26358. <a href="https://doi.org/10.1371/journal.pone.0026358">https://doi.org/10.1371/journal.pone.0026358</a>
- Fluge, O., Risa, K., Lunde, S., Alme, K., Rekeland, I. G., Sapkota, D., Kristoffersen, E. K., Sorland, K., Bruland, O., Dahl, O., & Mella, O. (2015). B-Lymphocyte Depletion in Myalgic Encephalopathy/ Chronic Fatigue Syndrome. An Open-Label Phase II Study with Rituximab Maintenance Treatment. *PLoS One*, *10*(7), e0129898. https://doi.org/10.1371/journal.pone.0129898
- Helmstaedter, C., Lendt, M., & Lux, S. (2001). Verbaler Lem-und Merkfähigkeitstest: VLMT; Manual. Beltz-test.
- Klok, F. A., Boon, G., Barco, S., Endres, M., Geelhoed, J. J. M., Knauss, S., Rezek, S. A., Spruit, M. A., Vehreschild, J., & Siegerink, B. (2020). The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. *Eur Respir J*, *56*(1). https://doi.org/10.1183/13993003.01494-2020
- Lenth, R. (2024). Emmeans: Estimated Marginal Means, Aka Least-Squares Means.
- Nasreddine, Z. S., Phillips, N. A., Bédirian, V., Charbonneau, S., Whitehead, V., Collin, I., Cummings, J. L., & Chertkow, H. (2005). The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. *J Am Geriatr Soc*, *53*(4), 695–699. https://doi.org/10.1111/j.1532-5415.2005.53221.x
- Reitan, R. M., & Wolfson, D. (1993). *The Halstead-Reitan neuropsychological test battery : theory and clinical interpretation* (2nd ed.). Neuropsychology Press.
- RUBIN, D. B. (1976). Inference and missing data. *Biometrika*, *63*(3), 581–592. https://doi.org/10.1093/biomet/63.3.581
- Scheibenbogen, C., Loebel, M., Freitag, H., Krueger, A., Bauer, S., Antelmann, M., Doehner, W., Scherbakov, N., Heidecke, H., Reinke, P., Volk, H. D., & Grabowski, P. (2018). Immunoadsorption to remove ss2 adrenergic receptor antibodies in Chronic Fatigue Syndrome CFS/ME. *PLoS One*, *13*(3), e0193672. https://doi.org/10.1371/journal.pone.0193672
- Schmidt, K., & Metzler, P. (1992). Wortschatztest (WST). Beltz Test GmbH. In: Weinheim.
- Sletten, D. M., Suarez, G. A., Low, P. A., Mandrekar, J., & Singer, W. (2012). COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. *Mayo Clin Proc*, 87(12), 1196–1201. https://doi.org/10.1016/j.mayocp.2012.10.013
- Strober, L. B., Bruce, J. M., Arnett, P. A., Alschuler, K. N., Lebkuecher, A., Di Benedetto, M., Cozart, J., Thelen, J., Guty, E., & Roman, C. (2020). A new look at an old test: Normative data of the symbol digit modalities test -Oral version. *Mult Scler Relat Disord*, *43*, 102154. https://doi.org/10.1016/j.msard.2020.102154
- Sturm, W., Willmes, K., & Horn, W. (2015). LPS 50: Leistungsprüfsystem für 50-bis 90-Jährige. In: Hogrefe.
- Tölle, M., Freitag, H., Antelmann, M., Hartwig, J., Schuchardt, M., van der Giet, M., Eckardt, K. U., Grabowski, P., & Scheibenbogen, C. (2020). Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Efficacy of Repeat Immunoadsorption. *J Clin Med*, *9*(8). https://doi.org/10.3390/jcm9082443
- van Buuren, S., & Groothuis-Oudshoom, K. (2011). mice: Multivariate Imputation by Chained Equations in R. *Journal of Statistical Software*, *45*(3), 1 67. https://doi.org/10.18637/jss.v045.i03
- Van Buuren, S., & Van Buuren, S. (2012). Flexible imputation of missing data (Vol. 10). CRC press Boca Raton, FL.
- Ware, J. E., Jr., & Sherbourne, C. D. (1992). The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. *Med Care*, *30*(6), 473–483.
- Wechsler, D. (2008). Wechsler adult intelligence scale (WAIS-IV). Pearson, The Psychological Corporation.

Yang, M., Keller, S., & Lin, J. S. (2019). Psychometric properties of the PROMIS((R)) Fatigue Short Form 7a among adults with myalgic encephalomyelitis/chronic fatigue syndrome. *Qual Life Res*, 28(12), 3375–3384. <a href="https://doi.org/10.1007/s11136-019-02289-4">https://doi.org/10.1007/s11136-019-02289-4</a>
Zimmermann, P., & Fimm, B. (2004). Kapitel 10 Die Testbatterie zur Aufmerksamkeitsprüfung (TAP).

Diagnostik von Konzentration und Aufmerksamkeit, 177.

14 Appendices

## 14.1 Flow Chart

# **CONSORT 2010 Flow Diagram**



# 14.2 Planned tables sample

Table 14.2.1 Baseline characteristics

| | In total | Intervention | Control |
|---|---|---|---|
| Baseline characteristics | (n=) | group<br>(n=) | group<br>(n=) |
| Age at randomization (years) | | () | () |
| Mean (SD), Median (IQR), [Min, Max] | | | |
| <b>Sex</b> , n <sub>.</sub> (%) | | | |
| male | | | |
| female | | | |
| diverse | | | |
| Ethnicity, n (%) | | | |
| Caucasian | | | |
| African | | | |
| Asian | | | |
| Other | | | |
| Unknown | | | |
| BMI (kg/m²), Mean (SD), Median (IQR), [Min, | | | |
| Max] | | | |
| Education, n (%) | | | |
| No school-leaving certificate, | | | |
| lower secondary school leaving certificate | | | |
| (Hauptschule), | | | |
| higher secondary school leaving certificate | | | |
| (Realschule), | | | |
| grammar school (Gymnasium), | | | |
| completed vocational training, | | | |
| degree of a university of applied sciences, | | | |
| University, | | | |
| Unknown | | | |
| Employment status, n (%) | | | |
| employed | | | |
| self-employed | | | |
| currently unable to work pension | | | |
| student | | | |
| unknown | | | |
| Pre-existing Comorbidities, n (%) | | | |
| Diseases of the circulatory system | | | |
| Diseases of the urogenital system | | | |
| Diseases of the genitourinary system | | | |
| Diseases of the digestive system Endocrine, Diseases of the | | | |
| musculoskeletal system and | | | |
| connective tissue | | | |
| Endocrine, nutritional and | | | |
| metabolic diseases | | | |
| Injuries, Poisoning and | | | |
| certain other consequences of external | | | |
| causes | | | |
| Smaking status n (9/) | | | |
| Smoking status, n (%) Current smoker | | | |
| Canoni dinokoi | | | |

former smoker never smoker unknown

Known allergies, n (%)

SARS-Cov-2 diagnosis in connection to fatigue,  $n \ (\%)$ 

Other infection in connection to fatigue, n (%)

Time from fatigue onset to study inclusion in days, Mean (SD), Median (IQR), [Min, Max]

Table 14.2.2 primary and secondary outcomes descriptive tables (examples)

| | Intervention<br>group<br>(n=) | Control<br>group<br>(n=) |
|---|---|---|
| Chalder Fatigue score, Mean (SD), Median | | |
| (IQR), [Min, Max] | | |
| baseline | | |
| EOT | | |
| 1 month | | |
| 4 months | | |
| 6 months | | |
| PCFS Scale, Mean (SD), Median (IQR), [Min, | | |
| Max] | | |
| Baseline | | |
| 1 month | | |
| 2 months | | |
| 4 months | | |
| 6 months | | |
| SF 36 physical domain, Mean (SD), Median (IQR), [Min, Max] | | |
| Baseline | | |
| 1 month | | |
| 2 months | | |
| 4 months | | |
| 6 months | | |

Table 14.2.3 Primary endpoint - Chalder Fatigue score after 2 months

| Study group | Chalder Fatigue score after 2<br>months<br>mean (95% CI) | Mean difference<br>(Intervention – Control)<br>(95% CI) | p-value |
|---|---|---|---|
| Intervention | | | |
| Control | | | |

Table 14.2.4 Secondary endpoints (examples)

| EORTC | Mean | (95%CI) | Mean difference | p- |
|---|---|---|---|---|
| | Intervention group (IG) | Control group (CG) | (IG – KG)<br>(95% CI) | values |
| Chalder Fatigue score | | | | |
| EOT | | | | |
| 1 month | | | | |
| 4 months | | | | |
| 6 months | | | | |
| PCFS Scale | | | | |
| 1 month | | | | |
| 2 months | | | | |
| 4 months | | | | |
| 6 months | | | | |
| SF 36 physical domain | | | | |
| 1 month | | | | |
| 2 months | | | | |
| 4 months | | | | |
| 6 months | | | | |

# 14.3 Planned listings sample for AEs SAEs

| Patient ID | Treatment<br>Arm | Age at baseline | Sex | Resolution<br>Date (YYYY-<br>MM-DD) | Duration<br>(Days) | Severity | Causality | Action<br>Taken | Outcome |
|---|---|---|---|---|---|---|---|---|---|

\_\_\_\_\_

# 14.4 Planned graphics sample

Figure 1: Chalder Fatigue scale over time, simulated data (n=44 intervention group, n=22 control group)



Figure 2: effect estimates for intervention for Chalder Fatigue Scale (n=44 in intervention group, n=22 in control group), (simulated data)



